CLINICAL TRIAL: NCT02372214
Title: Impact of a Patient-specific Simulation on the Learning Curve of Infra-renal Aneurysm Endovascular Repair
Brief Title: Production of a Patient-specific Simulator for Endovascular Aneurysm Repair Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3Daneurysm
Record Dates: First submitted 2015-02-02; First posted 2015-02-26 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2016-07

CONDITIONS: Aneurysm
Keywords: Endovascular Procedures; 3D printing; Simulation; Training; Learning curve; Education
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (No Intervention): 30 patients/5 vascular surgery residents The residents of the last year of vascular surgery will perform the procedure under supervision of a senior surgeon
- Group 2 (Experimental): 30 patients/5 vascular surgery residents Patients will have their aneurysm impressed by a 3D printing. The senior vascular surgeon and the residents of this group will be able to practice the procedure in the model as many times as they wish before the surgery. After the training, the EVAR will be performed according to the routine of the hospital.
  Interventions: Procedure: Training

INTERVENTIONS:
Procedure: Training — Patients will have their aneurysm impressed by a 3D printing. The senior vascular surgeon and the residents of this group will be able to practice the procedure in the model as many times as they wish before the surgery. After the training, the EVAR will be performed according to the routine of the hospital.
  Arms: Group 2

SUMMARY:
The purpose of this study is to produce a patient-specific simulator for endovascular infra-renal aneurysm repair training and than analyze the effect of simulator training on the performance of vascular surgery residents.

DETAILED DESCRIPTION:
Title: Production of a patient-specific simulator for endovascular aneurysm repair training.

Clinics Hospital of São Paulo University Medical School

Introduction

The aorta aneurysm is a common clinical condition that implies in considerable threatening to the life of patients. Before the year 2000, 99% of the abdominal aortic aneurysm (AAA) repair where performed with open surgery. Nevertheless, Catheter-based minimally invasive interventions are rapidly becoming the preferred initial treatment in patients with vascular disease . After 2004, the endovascular treatment of AAA increased to 52%. This changing venue requires a shift in our approach to training both fellows as well as general surgical residents during their exposure to vascular surgery.

Currently, supervised training with progressive exposure to procedures is the norm. Nevertheless, simulations based training may allow a shortening of the learning curve and avoid the exposure of the patients to unnecessary risks.

Using the rapid prototyping it is possible to build models in flexible materials that are helpful for training surgeons while simulating surgical procedures in a very realistic manner.

The possibility of training surgical procedures in general as well as patient-specific procedures might improve the surgeon's abilities and results . Rapid prototyping models allow for intensive training of young surgeons, e.g., for endovascular stent implantation simulating in vivo conditions and real tissues without any risk of patient complications and with no exposure of the surgeon to radiation or biologic risks.

After being adequately trained on models, surgeons feel more confident while going to the operating room for actual surgery. Besides, the pre-operative simulation of a specific and complex surgery provides a unique opportunity to employ surgical steps in order to determine the best operating strategy.

Simulators for catheter-based intervention have been available for approximately 5 years, and the technology is evolving rapidly. Currently, simulators are expensive and access has been limited. The ultimate test of simulation is to demonstrate that performance improves in the operating room.

To this end, we designed a randomized prospective study to describe the creation of a patient-specific simulator for training in endovascular infra-renal aneurysm correction and we will analyze the effect of simulator training on the performance of vascular surgery residents.

Objectives:

Primary: Production of a patient-specific simulator for training in endovascular infra-renal aneurysm repair.

Secondary: Analyze the effect of simulator training on the performance of vascular surgery residents.

Methods:

Production of a patient-specific simulator: The process chain on the production of a three-dimensional rapid prototype model consists of the following three steps: Image acquisition, Image post-processing and 3D printing. Patients will undergo a angioCT, with slice thickness of 1mm. Acquired data will be saved in the common DICOM format (Digital Imaging and Communications in Medicine). Dedicated high performance workstations equipped with post-processing tools will be used for processing the DICOM images generated during acquisition. The DICOM data will be transformed into a STL (Surface Tesselation Language) file format. The 3D machine reads in data from a CAD drawing and lays down successive layers of liquid, powder, or the sheet material, and in this way builds up the model from a series of cross sections. With that, a patient-specific pulsatile model will be produced.

Analyze the effect of simulator training on the performance of vascular surgery residents: The study will be performed during a period of two years (2014 and 2015), at the Clinics Hospital of São Paulo University Medical School.

All the endovascular aneurysm repair (EVAR) performed in during this time will be analyzed. According to the average number of EVAR in this service, we calculate that this research will include at least 60 patients.

Ten vascular surgery residents coursing the last year of practice will be randomized into the 2 groups (this is the total number of residents in our service).

Inclusion Criteria:

* Patients with infra-renal aneurysm with diameter of 5,5cm or more
* Residents of the last year of vascular surgery at Clinics Hospital of São Paulo University Medical School

Exclusion Criteria:

* Patients not suitable for endovascular aneurysm repair
* Patients with iliac aneurysm that require iliac bifurcated grafts
* Residents who don't want participate

  * Group 1 (30 patients/5residents): patients will undergo endovascular aneurysm repair according to the hospital routine. The residents will perform the procedure under supervision of a senior surgeon. It is an observational part of the study, which has already been done during the year 2014.
  * Group 2 (30 patients/5residents): patients will have their aneurysm impressed by a 3D printing. The senior vascular surgeon and the residents of this group will be able to practice the procedure in the model as many times as they wish before the surgery. After the training, the EVAR will be performed according to the routine of the hospital.

During the surgery, objective parameters will be analyzed: radioscopy time, volume of contrast injected, total procedure time, number of catheters and guide-wires used, technical success. The patients will be followed until they leave the hospital. Morbidity (myocardial infarction, renal failure, pulmonary complications) and mortality during the peri-operative time (30 days) will be analyzed. The surgeon will answer a questionnaire about the experience. The data from the two groups will be compared.

This study is approved by the national ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients with infra-renal aneurysm with diameter of 5,5cm or more
* Residents of the last year of vascular surgery at Clinics Hospital of São Paulo University Medical School

Exclusion Criteria:

* Patients not suitable for endovascular aneurysm repair
* Patients with iliac aneurysm that require iliac bifurcated grafts
* Residents who don't want participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Fluoroscopy time | 2 years - all the surgeries
  The total fluoroscopy time in every surgery will be counted, measured in minutes

SECONDARY OUTCOMES:
Number of participants with Myocardial infarction. | 30 days
  The Number of participants with Myocardial infarction (CKMB or Troponin positive curve or change in ECG) within 30 days of the surgery.
Number of participants with Renal disfunction | 30 days
  Number of participants with renal disfunction (necessity of hemodialysis or enhance of creatinine level) within 30 days of the surgery.
Death | 30 days
Number of participants with Pulmonary complications | 30 days
  Number of participants with Pulmonary complications (Pneumonia, Pulmonary congestion) within 30 days of the surgery.
Technical success (Endoprosthesis located in the right position, no endoleak type 1) | 30 days
  Endoprosthesis located in the right position, no endoleak type 1
Contrast volume in each surgery | 2 years
  The volume of contrast used in all the surgeries will be measured in milliliters during the period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson De Luccia, PhD, Study Director — Professor of São Paulo University Medical School
Locations (1):
- Clinics Hospital of São Paulo University Medical School, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided